CLINICAL TRIAL: NCT04746950
Title: ALICIA (Observational Prospective Study of Acalabrutinib in CLL Therapy in Real Clinical Practice in Russia)
Brief Title: ALICIA (Acalabrutinib in CLL Therapy)
Acronym: ALICIA
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00021
Record Dates: First submitted 2020-12-23; First posted 2021-02-10 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
This is a multicenter non-interventional observational study conducted with a single hand arm to collect real-world data. In this study, commercially available acalabrutinib will be used as prescribed treatment for CLL as per the treating physician's best clinical judgement. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

A multi-center collaborative effort in 15 centers selected from regions within Russia will help capture more patients into the database, rather than limiting the data to a single institution. This will be critical for:

* increasing database sample size
* reducing bias (single institution bias)
* increasing result's generalizability to the whole Russian population Being an observational study, only data available from routine clinical practice and standard of care (SoC), in line with national and international laws and regulations, will be recorded.

Patients will be treated according to prescribing information, with visit frequency and assessments performed according to routine medical practice and SoC. Only data corresponding to these visits and assessments will be collected as part of the study.

Data for the study will be transcribed and entered into an electronic Case Report Form (eCRF) from the patient's medical records. The site investigator will be responsible for ensuring that all required data is collected and entered into the eCRF with the involvement of clinical research organization

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed diagnosis of CLL
* Patient started treatment with monotherapy acalabrutinib (prescribed by physician decision no more than 4 weeks ago before screening)
* Capability of providing written Informed Consent Form

Exclusion Criteria:

* Patients not corresponded to inclusion criteria
* Pregnancy
* Lactation
* Patients included in open-label trials
* Previous Bruton tyrosine kinase inhibitors (BTKI) treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Enrolled set will be represented by eligible patients who have signed an informed consent form to participate in the study.
  It is estimated that approximately 200 patients will be enrolled in the study. Study population will consist of adult patients with diagnosed CLL ≥ 18 years old (treatment naïve (TN) or relapsed/refractory (R/R)) for whom acalabrutinib in monotherapy was prescribed by treating physician decision no more than 4 weeks ago before screening.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
• progression-free survival (rwPFS) in patients with CLL who are treated with acalabrutinib in clinical practice in Russia | Up to 2 years
• incidence of adverse events and serious adverse events in CLL patients treated with acalabrutinib in clinical practice in Russia | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - Research Site, Ufa, Bashkortostan Republic
  - Research Site, Kaliningrad, Kaliningrad Oblast
  - Research Site, Khabarovsk, Khabarovskiy Kray
  - Research Site, Syktyvkar, Komi
  - Research Site, Krasnoyarsk, Krasnoyarsk Region
  - Research Site, Saint Petersburg, Leningradskaya Oblast'
  - Research Site, Moscow, Moscow Oblast
  - Research Site, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Research Site, Novosibirsk, Novosibirsk Oblast
  - Research Site, Yakutsk, Sakha Republic
  - Research Site, Saratov, Saratov Oblast

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home